CLINICAL TRIAL: NCT01963858
Title: Effect of Functional Relaxation on Patients Undergoing Colonoscopy: A Prospective Randomized Controlled Trial
Brief Title: Effect of Functional Relaxation on Patients Undergoing Colonoscopy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Catholic University of Korea (Other)
Responsible Party: Principal Investigator, Jeong-Seon Ji, MD, PhD, The Catholic University of Korea
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: Relaxation
Record Dates: First submitted 2013-10-12; First posted 2013-10-16 (Estimated); Last update posted 2016-09-21 (Estimated); Status verified 2016-09

CONDITIONS: Colonoscopy; Relaxation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Functional relaxation (Experimental): Functional relaxation
  Interventions: Procedure: Functional relaxation
- No relaxation (Active Comparator): No relaxation
  Interventions: Procedure: No relaxation

INTERVENTIONS:
Procedure: Functional relaxation — Functional relaxation during colonoscopy
  Arms: Functional relaxation
Procedure: No relaxation — No relaxation during colonoscopy
  Arms: No relaxation

SUMMARY:
Patient attending for colonoscopy are generally worried and anxious. Fear of discomfort is the most common reason for low acceptance of colonoscopy. Several methods have been used to minimize patient discomfort, including the use of paediatric colonoscopes, variable stiffness colonoscopes, gastroscopes, music, audio distraction, or simply allowing the patients to participate in administration of medication. Although a potential benefit from some of these methods has been suggested, no clear recommendations have been made so far. We hypothesized functional relaxation reduces discomfort during colonoscopy.

ELIGIBILITY:
Inclusion Criteria:

* Patient undergoing screening or surveillance colonoscopy

Exclusion Criteria:

* Previous colorectal resection

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2013-10; Primary Completion 2016-04 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Patient's abdominal pain during colonoscopy | 1 day

SECONDARY OUTCOMES:
Patient satisfaction | 1 day

OTHER OUTCOMES:
State Trait Anxiety Inventory (STAI) | 1 day

CONTACTS AND LOCATIONS:
Locations (2):
- South Korea (2):
  - Incheon St. Mary's hospital, Catholic university of Korea, Incheon
  - Uijeongbu St. Mary's Hospital, The Catholic University of Korea, Uijeongbu-si

IPD SHARING:
Plan to Share IPD: No